CLINICAL TRIAL: NCT04881903
Title: Developing a Mobile Intervention to Reduce Suicidal Cognitions in Veterans (COR 19-490)
Brief Title: Developing a Mobile Intervention to Reduce Suicidal Cognitions in Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRX 21-001
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Suicide
Keywords: Suicide; Suicide cognitions; Anger; Mobile intervention
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: Participants will use the Mobile Intervention for Suicidal Thoughts (MIST) intervention for 4 weeks, followed by the Mobile Intervention for Reducing Anger (MIRA) for another 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MIST intervention followed by MIRA intervention (Experimental): These are both mobile interventions that use interpretation bias modification (IBM) techniques to reduce cognitive biases. The MIST app targets suicidal cognitions and the MIRA app targets hostile interpretation bias (which contributes to anger). The MIRA application has already been developed, but the MIST application is newly developed based on the same procedures. All participants will complete the MIST intervention and provide feedback so that we can refine it. We will also be collecting EMA data on to examine how changes to suicide cognitions and hostile interpretation bias (by use of the two apps) affects suicidal ideation and functioning.
  Interventions: Behavioral: Mobile Intervention for Suicidal Thoughts (MIST); Behavioral: Mobile Intervention for Reducing Anger (MIRA)

INTERVENTIONS:
Behavioral: Mobile Intervention for Suicidal Thoughts (MIST) — This is an interpretation bias modification intervention that is designed to target cognitive factors that contribute to suicide risk. Participants will be instructed to complete at least 5 treatment sessions per week for a period of 4 weeks. Each session takes approximately 10 minutes.
Behavioral: Mobile Intervention for Reducing Anger (MIRA) — This is an interpretation bias modification intervention that is designed to target hostile interpretation bias. Participants will be instructed to complete at least 5 treatment sessions per week for a period of 4 weeks. Each session takes approximately 10 minutes.

SUMMARY:
Suicide cognitions are conceptualized as enduring, chronic vulnerability factors that predispose individuals to suicidal crises. Therefore, modification of these beliefs may reduce suicidal thoughts and behaviors. The goal of this research is to develop, refine, and pilot-test a mobile intervention to reduce cognitions that contribute to elevated suicide risk and to assess the impact of reductions in suicide cognitions and anger cognitions on suicide risk and functioning.

DETAILED DESCRIPTION:
Suicide cognitions are conceptualized as enduring, chronic vulnerability factors that predispose individuals to suicidal crises. Therefore, modification of these beliefs may reduce suicidal thoughts and behaviors. In addition to suicide cognitions, another potentially modifiable risk factor for suicide is anger. The goal of this research is to develop, refine, and pilot-test a mobile interpretation bias modification intervention to reduce cognitions that contribute to elevated suicide risk and to assess the impact of reductions in suicide cognitions and hostile interpretation bias (a cognitive bias that is associated with anger) on suicide risk and functioning.

ELIGIBILITY:
Inclusion Criteria:

* Veterans 18 years or older
* Diagnosed with PTSD, established via the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5)
* Report a score of 12 on the 5-item Dimensions of Anger Reactions Scale
* Can read at least 6th grade level material
* Report a score of 1-3 (indicating ideation without intent) on the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Have attended a mental health appointment within the past month, with another scheduled in the following month (i.e., be engaged in treatment with a mental health provider)

Exclusion Criteria:

* Diagnosed with bipolar or psychotic disorder.
* Current substance use disorder.
* Current imminent suicide risk or homicidal ideation requiring immediate intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten H Dillon, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MIST Intervention Followed by MIRA Intervention
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MIST Intervention Followed by MIRA Intervention
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 4
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Recruited
Description: Participant feasibility expectation will be met if recruitment is 75% (i.e., N = 8) or greater of recruitment expectation (N = 10).
Time Frame: Through study completion (approximately 10 months)
Measure: Count of Participants; unit: Participants
Arm/Group | MIST Intervention Followed by MIRA Intervention
Number analyzed (Participants) | 10
Participants | 10

2. Primary Outcome: Number of Enrolled Participants Who Complete the MIST Intervention
Description: Treatment retention feasibility goal will be met if attrition from the MIST intervention is no more than 25% (i.e., not more than 3).
Time Frame: Post-MIST assessment visit (approximately one month after enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | MIST Intervention Followed by MIRA Intervention
Number analyzed (Participants) | 10
Participants | 10

3. Primary Outcome: Number of Participants Reporting Satisfaction With MIST App: Client Satisfaction Questionnaire
Description: Patient satisfaction will be assessed with item #7 from the Client Satisfaction Questionnaire. This item is scored on a scale of 1 to 4, with one indicating lower satisfaction and 4 indicating greater satisfaction. The patient satisfaction goal will be met if 80% or greater of participants indicate score a 3 or 4 on this item (i.e., at least 8 participants score a 3 or 4).
Time Frame: Post-MIST assessment visit (approximately one month after enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | MIST Intervention Followed by MIRA Intervention
Number analyzed (Participants) | 10
Participants | 8

4. Primary Outcome: MIST App Utilization
Description: MIST app utilization goal will be met if MIST app utilization rates are greater than 50% of expected use (i.e., mean # of sessions completed is greater than 10).
Time Frame: Post-MIST assessment visit (approximately one month after enrollment)
Measure: Mean (Standard Deviation); unit: treatment sessions completed
Arm/Group | MIST Intervention Followed by MIRA Intervention
Number analyzed (Participants) | 10
treatment sessions completed | 15.30 (4.35)

ADVERSE EVENTS:
Time Frame: 2.5 months
Description: No adverse events occurred during the MIRA or MIST interventions; all adverse events occurred during the screen portion of the study.
Groups:
- MIST Intervention: Mobile Intervention for Suicidal Thoughts (MIST): This is an interpretation bias modification intervention that is designed to target cognitive factors that contribute to suicide risk. Participants will be instructed to complete at least 5 treatment sessions per week for a period of 4 weeks. Each session takes approximately 10 minutes.
- MIRA Intervention: Mobile Intervention for Reducing Anger (MIRA): This is an interpretation bias modification intervention that is designed to target hostile interpretation bias. Participants will be instructed to complete at least 5 treatment sessions per week for a period of 4 weeks. Each session takes approximately 10 minutes.
- Screening: This is the period between consent and beginning the intervention.
Arm/Group | MIST Intervention | MIRA Intervention | Screening
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIST Intervention (N=10) | MIRA Intervention (N=10) | Screening (N=10)
Distress during screen (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) — Temporary distress related to completing self-report measures about trauma and/or structured interviews about trauma and posttraumatic stress disorder symptoms.
Frustration with dealing with virtual visit platform (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT04881903/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT04881903/ICF_001.pdf